CLINICAL TRIAL: NCT00736554
Title: Prevalence of MRSA in Skin and Soft Tissue Infections in Two Ontario Emergency Departments.
Brief Title: What is the Prevalence of Methicillin-Resistant Staphylococcus Aureus in Skin and Soft Tissue Infections Presenting to the Emergency Departments of a Canadian Academic Health Care Center?
Acronym: CA-MRSA
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Dr. Christopher Fernandes, London Health Sciences Centre
Other Study IDs: R-08-173; 13871E (Other: REB)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Bacterial Infections; Gram-Positive Bacterial Infections; Staphylococcal Infections
Keywords: Staphylococcus aureus; CA-MRSA; skin and soft tissue infections; resistance; emergency department
MeSH Terms: conditions — Bacterial Infections; Gram-Positive Bacterial Infections; Staphylococcal Infections; Soft Tissue Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Staphylococcus aureus is the most common bacteria responsible for skin, bone, and muscle infections. Recent studies from the United States have suggested that a type of this bacterium called methicillin resistant S. aureus (MRSA) has become dramatically more common, especially the community strain. However, Canadian data is still largely lacking. This study aims to determine the prevalence of community acquired (CA) MRSA among patients presenting with skin and soft tissue infections to the Urgent Care Center and Emergency Departments in London, Ontario. This will be determined by taking swabs at enrollment from patient's noses, throats, and sites of infection. Patients will be asked to complete a health questionnaire with the goal of identifying risk factors associated with CA-MRSA. Through follow-up swabs of participants' noses and throats at one and three months, the effects of treatment on patient's carrying MRSA will be determined. Results may be used to form guidelines for empirical S aureus treatment in the region, reducing possible morbidity and mortality from delayed or suboptimal treatment of CA-MRSA infections. Improved understanding of risk factors associated with MRSA infection in a Canadian setting, may also change the practice of physicians considering empiric antibiotic therapy for skin and soft tissue infections.

DETAILED DESCRIPTION:
Objective & Hypothesis: The objective of this prospective study is to determine the prevalence of MRSA and community acquired MRSA (CA-MRSA) in adult patients (>17yrs old) presenting with skin or soft tissue infections to the emergency departments (EDs) of an academic health care setting in London, Ontario. Secondary objectives will include the identification of demographic and clinical variables associated with MRSA, characterization of MRSA antimicrobial susceptibilities and genotypes, and determining the effects of treatment on MRSA colonization. We believe that the prevalence of MRSA and CA-MRSA in London, Ontario will be lower than rates recently published by academic hospitals from the United States. The hypothesis of the study is that patients presenting to the Emergency Departments in London, Ontario with skin and soft tissue infections will have a 10% prevalence of CA-MRSA, but certainly the prevalence may be much higher.

Purpose: Results from this research may be used as part of the guidelines for empirical S aureus treatment in the region, thus reducing possible morbidity and mortality from delayed or suboptimal treatment of CA-MRSA infections. This information, along with an improved understanding of risk factors associated with MRSA infection in a Canadian setting, has the potential to change the practice of physicians who are considering empiric antibiotic therapy for skin and soft tissue infections.

This study will focus on the epidemiology of patients with skin or soft tissue infections presenting to the adult emergency departments (EDs) at the London Health Sciences Centre (LHSC) and the Urgent Care Center at St. Joseph's Health Centre (SJHC). By using a comparison group of non CA-MRSA infections, the proportion of CA-MRSA with relation to the total MRSA and methicillin sensitive Staphylococcus aureus (MSSA) in the region will be investigated. The study will also investigate the risk factors in the CA-MRSA population including: demographics, housing history, contact with the health care system, past CA-MRSA infection, asymptomatic CA-MRSA colonization, colonization/infection of close contacts, involvement in contact sports/team sports, hygienic body shaving, chronic skin disorders, recurrent/recent antibiotic use, IV drug use, contact with incarcerated individuals, and chronic disease.

Through follow-up visits at one and three months involving nares and throat swabs of patients initially testing positive for MRSA the effects of treatment on MRSA colonization will be determined. Furthermore, a follow-up questionnaire will be administered to all patients at one month to determine complication rates for patients colonized with MRSA versus those not colonized.

The current recommendations for antibiotic treatment of unknown S. aureus infection are based on clinical judgment, and therefore an understanding of regional incidence and susceptibility of CA-MRSA are essential for empiric treatment. Through the microbiological analysis of the cases, laboratory parameters and antibiotic susceptibility of CA-MRSA presenting to LHSC will be established. As well, the clinical characteristics of these patients will be documented to aid clinicians in recognizing patients presenting with CA-MRSA.

Experimental Design: This study will be a prospective prevalence study involving adult patients (>17years old) with skin and soft-tissue infections presenting to the Emergency Departments of LHSC (University Hospital and Victoria Hospital) as well as to the Urgent Care of SJHC. These departments have a combined approximate total of 150,000 visits per year. The study has an expected enrollment of 152 patients from July 2008- July 2009. The study will continue until three months after the last patient has been enrolled so that follow-up nasal and throat swabs may be obtained, if applicable.

n = Z2 P (1-P) / d2 n = 1.962 * .10 (1- .10) / 0.052 n = 3.8416 * .10 * .90 / .0025 n = 138

While the investigators do not anticipate a problem with non-response or missing values, to take this into consideration, we will over-sample the above sample size by 10%. Therefore, we will recruit at least 152 patients to the study. Therefore, assuming 80% power, an estimated prevalence of 10%, and a precision level of 5%, 152 patients are needed to be 95% confident that the true proportion of MRSA in adult patients (>17yrs old) presenting with skin or soft tissue infections will be between 5% and 15%.

Written, informed consent will be obtained from all patients that meet the study inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (> 17 years) whose chief complaint is consistent with skin or soft tissue infection (cellulitis, necrotizing soft tissue infection, wound infection, ulcer, septic bursitis, abscess including furuncle/carbuncle/superficial skin abscess, paronychia, hordeolum, pilonidal abscess, acute lymphadenitis, pilonidal cyst without abscess, and impetigo).

Exclusion Criteria:

* Patients will be excluded if they refuse to participate or written, informed consent is not obtained.
* Additionally, patients with Bartholin cysts, odontogenic infections and perianal abscesses will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selection of Participants: The objective of this prospective study is to determine the prevalence of MRSA and community acquired MRSA (CA-MRSA) in adult patients (>17 yrs old) presenting with skin or soft tissue infections to the emergency departments (EDs) of an academic health care setting in London, Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher MB Fernandes, FRCP, FACEP, MD, Principal Investigator — The University of Western Ontario
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada